CLINICAL TRIAL: NCT01117181
Title: Apathy in Dementia Methylphenidate Trial (ADMET)
Acronym: ADMET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Medical University of South Carolina (Other); Johns Hopkins University (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AG033032-01 (NIH); R01AG033032-01 (NIH)
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Results first posted 2013-05-10 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Apathy; Alzheimer's Disease
Keywords: Alzheimer's disease; Apathy; Methylphenidate; Dopaminergic agents; Apathy Evaluation Scale; Dementia
MeSH Terms: conditions — Lethargy; Alzheimer Disease; Dementia | interventions — Methylphenidate; Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Experimental): Methylphenidate, target dose 20 mg per day (range 10-20 mg per day) and psychosocial intervention
  Interventions: Drug: Methylphenidate; Other: Psychosocial intervention
- Placebo (Placebo Comparator): matching placebo and psychosocial intervention
  Interventions: Drug: placebo; Other: Psychosocial intervention

INTERVENTIONS:
Drug: Methylphenidate — The target dose is 20 mg per day provided as two 10 mg doses administered orally. Patients will start by taking 10 mg daily (two 5 mg over-encapsulated tablets) for three days, at which time the dose will be increased to 20 mg per day (four 5 mg over-encapsulated tablets). In the event of significant side-effects, the dose will be reduced to a minimum of 10 mg per day. The study drug will be administered for 6 weeks.
  Other Names: Ritalin
  Arms: Methylphenidate
Drug: placebo — Patients will start with two capsules of placebo for three days, at which time the dose will be increased to four capsules. The dose may be reduced to a minimum of two capsules per day if there appears to be significant side-effects. Placebo will be administered for 6 weeks.
  Other Names: dummy pill
  Arms: Placebo
Other: Psychosocial intervention — The psychosocial intervention will consist of three components: a counseling session, the provision of education materials, and 24-hour availability for crises.
  The counseling session, in which a trained study clinician will counsel the primary caregiver, lasts approximately 20-30 minutes, and consists of the following elements:
  * Review and adjustment of the patient and caregiver supportive care plans
  * Emotional support and opportunity to ventilate feelings
  * Counseling regarding specific caregiving skills
  * Assistance with problem solving of specific issues that the caregiver brings to the sessions
  * Answers for questions regarding the educational materials
  The educational materials will consist of a copy of the book The 36-Hour Day

SUMMARY:
The Apathy in Dementia Methylphenidate Trial (ADMET) is a masked, placebo-controlled trial that will examine the efficacy and safety of methylphenidate for the treatment of clinically significant apathy in patients with Alzheimer's dementia.

DETAILED DESCRIPTION:
The Apathy in Dementia Methylphenidate Trial (ADMET), funded by the National Institute of Aging, is a Phase II, placebo-controlled, masked, 3-center randomized clinical trial. ADMET will enroll 60 patients with Alzheimer's disease (AD) and significant apathy from outpatient, nursing home, and assisted living facilities along with their primary caregiver. Eligible and willing patients will be randomly assigned to methylphenidate (20 mg per day) or placebo. At baseline and each in-person follow-up visit, all caregivers and patients will be provided with a standardized psychosocial intervention consisting of a counseling session, provision of educational materials, and 24-hour availability for crises. Efficacy and safety outcomes will be measured at baseline and at in-person follow-up visits at 2, 4, and 6 weeks following randomization. Telephone contact will take place at 1, 3, and 5 weeks after randomization.

ADMET has 80% power to detect a difference of at least 3.3 in change in the Apathy Evaluation Scale scores between the two treatment groups. It also has 80% power to detect an absolute difference of 35% or more in the change in the proportion of study participants improving on te Clinical Global Impression of Change, given that 20% to 305 of participants in the placebo group show improvement.

ELIGIBILITY:
Inclusion criteria:

* Possible or probable Alzheimer's disease (National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria), with Mini-Mental State Exam (MMSE) score of 10-26 inclusive; MMSE scores above 26 in those who nevertheless meet criteria for AD may be allowed with Steering Committee approval on a case by case basis
* Clinically significant apathy for at least four weeks for which either 1) the frequency of apathy as assessed by the Neuropsychiatric Inventory (NPI) is 'Very frequently', or 2) the frequency of apathy as assessed by the NPI is 'Frequently' or 'Often' AND the severity of apathy as assessed by the NPI is 'Moderate' or 'Marked'
* A medication for apathy is appropriate, in the opinion of the study physician
* Provision of informed consent for participation in the study by patient or surrogate (if the patient is unable to provide informed consent) and caregiver
* Availability of primary caregiver, who spends greater than ten hours a week with the patient and supervises his/her care, to accompany the patient to study visits and to participate in the study
* Sufficient fluency, of both the patient and caregiver, in written and spoken English to participate in study visits, physical exams, and outcome assessments
* No change to AD medications within the month preceding randomization, including starting, stopping, or dosage modifications
* Treatment with stable doses of selective serotonin reuptake inhibitor antidepressants(SSRIs) is appropriate if stable for 3 months prior to randomization. Other psychotropics(with the exclusion of antipsychotics), if stable for 3 months, may be allowed only with Steering Committee approval on a case by case basis.

Exclusion criteria:

* Meets criteria for Major Depressive Episode, by Diagnostic Statistical Manual of Mental Disorder - IV (TR) criteria
* Clinically significant agitation /aggression for which either 1) the frequency of agitation /aggression as assessed by the NPI is 'Very frequently', or 2) the frequency of agitation /aggression as assessed by the NPI is 'Frequently' AND the severity of the agitation as assessed by the NPI is 'Moderate', or 'Marked'
* Clinically significant delusions for which either 1) the frequency of delusions as assessed by the NPI is 'Very frequently', or 2) the frequency of delusions as assessed by the NPI is 'Frequently' AND the severity of the delusions as assessed by the NPI is 'Moderate', or 'Marked'
* Clinically significant hallucinations for which either 1) the frequency of hallucinations as assessed by the NPI is 'Very frequently', or 2) the frequency of hallucinations as assessed by the NPI is 'Frequently' AND the severity of the hallucinations as assessed by the NPI is 'Moderate', or 'Marked'
* Treatment with psychotropic medications in the 2 weeks prior to randomization with the exception of approved treatments for dementia (ChEIs and memantine), selective serotonin reuptake inhibitor antidepressants, and trazodone (if used as an aid to facilitate sleep and not as an antidepressant); other psychotropics (with the exclusion of antipsychotics), if stable for 3 months, may be allowed only with Steering Committee approval on a case by case basis. Note that antipsychotics are expressly prohibited.
* Treatment with methylphenidate is contraindicated in the opinion of the study physician
* Failure of treatment with methylphenidate in the past for apathy after convincing evidence of an adequate trial as judged by study physician
* Treatment with a medication that would prohibit the safe concurrent use of methylphenidate such as monoamine oxidase inhibitors and tricyclic antidepressants
* Need for acute psychiatric hospitalization or is suicidal
* Uncontrolled hypertension (medication non-compliance or past 3 months with a diastolic reading of 105 as verified by compartment pressure of the rectus sheath (CPRS))
* Symptomatic coronary artery disease deemed to be significant by study physician at the time of screening
* Lack of appetite that results in significant unintentional weight loss as determined by the study physician in the last three months
* Significant communicative impairments
* Current participation in a clinical trial or in any study that may add significant burden or affect study outcomes
* Hyperthyroidism, advanced arteriosclerosis, symptomatic cardiovascular disease, serious structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, or a family history of sudden death or death related to heart problems
* Glaucoma, pheochromocytoma, or known or suspected hypersensitivity to methylphenidate or its excipients
* Central Nervous System (CNS) abnormalities (e.g., cerebral aneurysm) and/or other vascular abnormalities such as vasculitis or pre-existing stroke, motor tics or a family history or diagnosis of Tourette's syndrome, seizures (convulsions, epilepsy), or abnormal EEGs
* Any condition that, in the opinion of the study physician, makes it medically inappropriate or risky for the patient to enroll in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Scherer, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; Jacobo Mintzer, MD, MBA, Study Chair — Medical University of South Carolina; Paul Rosenberg, MD, Principal Investigator — Johns Hopkins University; Krista Lanctot, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Medical University of South Carolina, Charleston, South Carolina
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Rosenberg PB, Lanctot KL, Drye LT, Herrmann N, Scherer RW, Bachman DL, Mintzer JE, ADMET Investigators. Safety and efficacy of methylphenidate for apathy in Alzheimer's disease: a randomized, placebo-controlled trial. J Clin Psychiatry. 2013 Aug;74(8):810-6. doi: 10.4088/JCP.12m08099. PMID 24021498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical center recruited from established outpatient clinics, from living facilities, by local physicians, and from targeted advertisements in local media. The recruitment period started June 2010 and ended October 2011.
Period: Overall Study
Arm/Group | Methylphenidate | Placebo
Started | 29 | 31
Completed | 28 | 29
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate | Placebo | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (8) | 75 (9) | 76 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41
  Canada | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Apathy Evaluation Scale (AES)
Description: Change in score of Apathy Evaluation Scale from baseline to 6 weeks; the minimum score is 18; the maximum score is 72. Higher scores indicate more severe apathy.
Time Frame: baseline to 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Methylphenidate: Methylphenidate, target dose 20 mg per day (range 10-20 mg per day), and psychosocial intervention
- Placebo: Placebo and psychosocial intervention
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 29 | 31
units on a scale | -1.9 (1.5) | 0.6 (1.4)

2. Primary Outcome: Alzheimer's Disease Cooperative Study- Clinical Global Impression of Change
Description: Proportion of individuals improving on Alzheimer's Disease Cooperative Study- Clinical Global Impression of Change (CGIC) from baseline to 6 weeks; the CGIC is a 7-point Likert scale used to rate each patient with the following scores: "marked worsening"(7), "moderate worsening" (6), "minimal worsening"(5), "no change"(4), "minimal improvement"(3), "moderate improvement"(2), "marked improvement"(1). Ratings were based on an interview with the caregiver and an examination of the patient. The CGIC requires the clinician to consider a number of aspects of apathy, such as level of initiative, level of interest, and emotional engagement.
Time Frame: baseline to 6 weeks
Measure: Number; unit: percentage of participants who improve
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 29 | 31
percentage of participants who improve | 21 | 3

3. Secondary Outcome: Digit Span
Description: Change in Digit Span from baseline to 6 weeks. The Wechsler Adult Intelligence Scale - Revised Digit Span is used to assess auditory attention and working memory. Both forward and backward span is assessed. Both tests consist of six number sequences that the psychometrist reads aloud one at a time. After each sequence is read, the participant must repeat the digits back in the same (forward) or reverse (backward) order. Scores range from 0 to 16, with higher numbers indicate better functioning.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 26 | 29
units on a scale | 0.46 (1.55) | -0.07 (1.25)

4. Secondary Outcome: Mini-Mental State Exam (MMSE)
Description: Change in Mini-Mental State Exam score from baseline to 6 weeks; this cognitive test estimates of dementia severity. Domains included orientation, memory, working memory, naming, following verbal and written commands, spontaneously writing a sentence, and copying two overlapping pentagons. The minimum MMSE score is 0; the maximum MMSE score is 30. Lower MMSE scores indicate more severe cognitive impairment.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 29 | 31
units on a scale | 1.3 (0.6) | -0.3 (0.6)

5. Secondary Outcome: Neuropsychiatric Inventory (NPI): Apathy Subscale
Description: Change from baseline to 6 weeks in neuropsychiatric symptoms in apathy subscore. Frequency (ranges from 1=occasionally, less than once/week to 4 = very frequently, once or more/day or continuously) and severity (1=mild, 2=moderate, 3=severe) scales are scored based on responses from an informed caregiver involved in the patient's life. To obtain the NPI score, the severity score is multiplied by the frequency score. Range is 0 to 12. Larger numbers indicate more severe behavioral disturbance.
Time Frame: baseline to week 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 29 | 31
units on a scale | -4.4 (0.6) | -2.6 (0.6)

6. Secondary Outcome: Vital Status
Description: vital status as measured by death
Time Frame: vital status at 6 weeks
Measure: Number; unit: participants who died
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 29 | 31
participants who died | 0 | 0

7. Secondary Outcome: Electrolytes
Description: Percent of participants with abnormal electrolyte values at 6 weeks as assessed by local laboratory
Time Frame: 6 weeks
Population: One patient in the active group completed all visit 6 assessments except for the blood collection for the electrolyte sample. This patient refused this procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 27 | 29
percentage of participants
  Sodium | 3.70 | 0
  Potassium | 14.81 | 10.34
  Chloride | 7.41 | 10.34
  Bicarbonate | 7.41 | 10.34

8. Secondary Outcome: Electrocardiogram (ECG)
Description: Abnormal electrocardiogram results at 6 weeks
Time Frame: 6 weeks
Measure: Number; unit: participants with abnormal ECG
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 29 | 31
participants with abnormal ECG | 20 | 15

ADVERSE EVENTS:
Time Frame: treatment period (i.e., 6 weeks)
Arm/Group | Methylphenidate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/31
Other Adverse Events (participants affected / at risk) | 29/29 | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate (N=29) | Placebo (N=31)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
drop in hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Methylphenidate (N=29) | Placebo (N=31)
agitation (Nervous system disorders) | 17 | 13/29
Anxiety (Nervous system disorders) | 17 | 10/29
weight loss (Metabolism and nutrition disorders) | 10 | 4/29 — greater than 2% at week 6
abdominal pain (Gastrointestinal disorders) | 6 | 4/29
Aggressive behavior or hostility (Psychiatric disorders) | 9 | 5/29
Angina (Cardiac disorders) | 2 | 1/29
Anorexia (Metabolism and nutrition disorders) | 6 | 5/29
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 14/29
Blood pressure changes (Vascular disorders) | 4 | 3/29
Blurry vision or eyesight changes (Eye disorders) | 0 | 3/29
Depressed appetite (Metabolism and nutrition disorders) | 8 | 7/29
Depressed mood (Psychiatric disorders) | 12 | 12/29
Distractibility (Social circumstances) | 11 | 8/29
Dizziness (Ear and labyrinth disorders) | 11 | 7/29
Drowsiness (General disorders) | 10 | 13/29
Dry mouth (Gastrointestinal disorders) | 7 | 6/29
Dyskinesia (Nervous system disorders) | 1 | 4/29
Hair loss (Endocrine disorders) | 2 | 1/29
Headache (General disorders) | 5 | 4/29
Hyperactivity (Nervous system disorders) | 5 | 1/29
Impaired learning (Social circumstances) | 4 | 7/29
Nausea (Gastrointestinal disorders) | 3 | 7/29
Skin rash, redness, or inflammation (Skin and subcutaneous tissue disorders) | 6 | 6/29
Tics (motor or verbal) (Nervous system disorders) | 0 | 4/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No